CLINICAL TRIAL: NCT00410189
Title: A Phase II, Open Label Study of ZD6474 in Previously Treated Subjects With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: BATTLE Program: ZD6474 in Previously Treated Subjects With NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0825
Record Dates: First submitted 2006-12-08; First posted 2006-12-12 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Lung Cancer
Keywords: Non-Small Cell Lung Cancer; NSCLC; Lung Cancer; ZD6474; Zactima; Vandetanib; BATTLE Program
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — vandetanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ZD6474 (Experimental): ZD6474 300 mg by mouth daily for 28 Days.
  Interventions: Drug: ZD6474

INTERVENTIONS:
Drug: ZD6474 — 300 mg by mouth daily for 28 Days.
  Other Names: Zactima; Vandetanib

SUMMARY:
Primary Objective:

* To determine the 8 week progression-free survival rate (i.e. disease control rate) in patients with advanced NSCLC who have failed at least one prior chemotherapy regimen.

Secondary Objectives:

* Determine the overall response rate
* Determine the overall survival
* Determine the time to disease progression
* Assess the safety/toxicity of the study treatment
* Assess biomarker modulation in the tumor tissue and serum samples from the treatment
* Assess plasma and intra-tumor concentrations of study treatment

DETAILED DESCRIPTION:
ZD6474 is designed to block the formation of new blood vessels. The growth of new blood vessels is called angiogenesis. Angiogenesis is thought to be important for the growth of tumors beyond a small size. Researchers want to find out if ZD6474 will limit new blood vessel growth in the tumor and "starve" the tumor by limiting blood flow to it.

In order to enroll in this study, you must also be enrolled in Protocol 2005-0823: A Biomarker-integrated study in Chemorefractory Patients with Advanced Non-Small Cell Lung Cancer. Protocol 2005-0823 is the screening study in a group of studies called the BATTLE program. Participants in Protocol 2005-0823 are assigned to one of the research studies. The results of your tumor analysis helped the study doctor determine to assign you to this particular treatment study.

While on study, you will take ZD6474 by mouth each morning. ZD6474 is swallowed as a whole tablet. The tablet should not be chewed, crushed, or divided and should be taken with 8 ounces of water and a small amount of food to lessen stomach discomfort. You should take ZD6474 at about the same time every day. Four (4) weeks is considered 1 treatment cycle. If you miss a dose and are unable to take the missed dose on the same day, you should take the next scheduled dose and the missed dose will not be made up. The dose of study medication may be repeated if vomiting occurs within 30 minutes of taking the study medication.

You will have routine blood tests (about 2 teaspoons) at Weeks 1, 2, 4, 8, 12, then every 4 weeks after that. You will have an electrocardiogram (ECG -- a test that measures the electrical activity of the heart) at Weeks 1, 2, 4, 8, 12, then every 3 months after that. Every 4 weeks, your complete medical history will be recorded and you will have a physical exam, including measurement of vital signs (blood pressure, heart rate, temperature, and breathing rate), a performance status evaluation, and weight. You will also have a routine urine test and your study doctor will ask you about any medications you are taking and your smoking history.

Every 2 cycles, your tumor will be evaluated by chest x-ray and computed tomography (CT) or magnetic resonance imaging (MRI) scans to evaluate the status of the disease. If you are taking coumadin, you will have blood drawn (about 1-2 teaspoons) to check your blood clotting function every week. You will be asked to bring your unused medication to each clinic visit.

You may continue receiving ZD6474 for as long as the cancer responds to study treatment. Your doctor may decide to take you off this study if you experience intolerable side effects, your medical condition gets worse, and/or you are unable to comply with study requirements. If you stop study treatment, you may be able to enroll in 1 of the remaining 3 protocols of the BATTLE program.

After you have stopped taking the study treatment, you will have a physical exam, including measurement of vital signs. Blood (about 2 teaspoons) and urine will be collected for routine tests. You will also have blood drawn (about 1-2 teaspoons) to check your blood clotting function. You will have a performance status evaluation, chest x-ray, ECG, and a CT or MRI scan. Following this evaluation, you will be contacted by telephone every 3 months for up to 3 years to see how you are doing.

You have the right to leave the study at any time. If you choose to stop participating in this study, you should contact the study chair and/or research nurse.

This is an investigational study. ZD6474 is an investigational drug that has been approved by the FDA for research use only. Up to 72 patients will take part in this multicenter study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a diagnosis of pathologically confirmed NSCLC by tumor biopsy and/or fine-needle aspiration.
2. The patient has a diagnosis of either stage IIIB, stage IV, or advanced, incurable NSCLC, and failed at least one front-line metastatic NSCLC chemotherapy regimen. (Patients who have failed adjuvant or locally advanced therapy within 6 months are also eligible to participate in study).
3. The patient has uni-dimensionally measurable NSCLC.
4. Karnofsky performance status >/= 60 or Eastern Cooperative Oncology Group (ECOG) performance status 0-2
5. The patient has biopsy accessible tumor.
6. The patient has adequate hematologic function as defined by an absolute neutrophil count (ANC) >/= 1,500/mm^3, platelet count >/= 100,000/mm^3, White Blood Count (WBC) >/= 3,000/ mm^3, and hemoglobin >/= 9 g/dL.
7. The patient has adequate hepatic function as defined by a total bilirubin level </= 1.5 times the upper limit of normal, and alkaline phosphatase, Alanine aminotranferease (ALT) or aspartate aminotransferase (AST) </= 2.5 times the upper limit of normal.
8. The patient has adequate renal function as defined by a serum creatinine level </= 1.5 mg/dL or a calculated creatinine clearance of >/= 60cc/minute.
9. The patient has prothrombin time (PT) < 1.5 times upper limit of normal
10. If patient has brain metastasis, they must have been stable (treated or asymptomatic) for at least 4 weeks after radiation if treated with radiation and not have used steroids for at least 1 week. Re-imaging performed after 2 weeks, upon completion of radiation therapy.
11. The patient is >/= 18 years of age.
12. The patient has signed informed consent.
13. The patient is eligible if disease free from a previously treated malignancy, other than a previous NSCLC, for greater than two years. Patients with a history of prior basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix are exempt from exclusion.
14. Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.Childbearing potential will be defined as women who have had menses within the past 12 months,who have not had tubal ligation or bilateral oophorectomy.Should a woman become pregnant or suspect that she is pregnant while participating in this study,she should inform her treating physician immediately.The patient,if a man,agrees to use effective contraception or abstinence.
15. Subject must be considered legally capable of providing his or her own consent for participation in this study.

Exclusion Criteria:

1. The patient has received prior investigational therapy, chemotherapy, surgery, or radiotherapy within 4 weeks of initiating study drug
2. The patient has undergone prior thoracic or abdominal surgery within 28 days of study entry, excluding prior diagnostic biopsy.
3. The patient has received radiation therapy to the measurable tumor within 6 months. Patients are allowed to have local irradiation for the management of tumor-related symptoms (bones, brain). However, if a patient has active new disease growing in the previously irradiated site, the patient will be eligible to participate in the study.
4. The patient has a significant medical history or unstable medical condition (unstable systemic disease: congestive heart failure (New York Heart Association Functional Classification class II or worse), recent myocardial infarction within 3 months, unstable angina, active infection (i.e. currently treated with antibiotics), uncontrolled hypertension). Patients with controlled diabetes will be allowed. Patient must be able to undergo procedure for tissue acquisition.
5. The patient has uncontrolled seizure disorder, active neurologic disease, or neuropathy >/= grade 2. Patients with meningeal or CNS involvement by tumor are eligible for the study if the above exclusion criteria are not met.
6. The patient is pregnant (confirmed by serum b-HCG if applicable) or is breastfeeding.
7. Any condition that is unstable or could jeopardize the safety of the patient and its compliance in the study, in the investigator's judgment
8. The patient is actively taking herbal remedies or over-the-counter biologics (e.g., shark cartilage, high dose antioxidants).
9. Patients will be allowed to have prior biologic (i.e. VEGF, EGFR, etc.) therapy. However, the patient will be excluded from a given study if he/she has received the same therapy as the clinical trial (i.e. If a patient has been previously treated with bevacizumab, they are allowed to enroll in any of the 4 studies. If a patient has been previously treated with erlotinib, they are excluded from the clinical trials with erlotinib). In addition, if a patient has been previously treated with gefitinib (Iressa), they are excluded from the clinical trials with erlotinib.
10. Patients must not have undergone minor surgery (e.g., central venous catheter placement) within 24 hours of treatment with ZD6474. Patients may not have undergone any major surgery (e.g. laparotomy, thoracotomy, or craniotomy) within four weeks of enrollment.
11. Patients may not have a history of a bleeding diathesis.
12. Significant cardiovascular event (e.g. myocardial infarction, superior vena cava syndrome (SVC), New York Heart Association (NYHA) classification of heart disease >/=2 within 3 months of entry of presence of cardiac disease that in the opinion of the investigator increases the risk of ventricular arrhythmia
13. History of clinically significant arrhythmia (multifocal PVCs, bigeminy, trigeminy, ventricular tachycardia), which is symptomatic or requires treatment (CTC grade 3) or a symptomatic sustained ventricular tachycardia. Atrial fibrillation, controlled on medication is not excluded.
14. Prior history of QT prolongation as a result from other medication that required discontinuation of that medication.
15. Congenital long QT syndrome or 1st degree relative with unexplained sudden death under 40 years of age.
16. QTc with Bazett's correction that is unmeasurable, or >/=480 msec on screening ECG. If a patient has QTc >/=480 msec on screening ECG, the screen ECG may be repeated twice (at least 24 hours apart). The average QTc from the three screening ECGs must be <480 msec in order for the patient to be eligible for the study). If the patient meets eligibility requirements in this way, the "baseline" QTc for this patient will be the average of the 3 ECGs (screen 1, screen 2, and pre-1st dose). Patients who are receiving a drug that has a risk of QTc prolongation are excluded if QTc is >/= 460 msec.
17. Any concomitant medications that affect QTc, induce Torsades de Pointes. (lists of relevant medications available that have a risk of Torsades de Pointes or QTc prolongation.) Drugs listed that in the investigator's opinion cannot be discontinued, are allowed however, must be monitored closely.
18. Potassium, calcium (ionized calcium or adjusted for albumin), or magnesium concentrations outside normal limits. Supplementation of electrolytes is permitted. Potassium level must be greater than or equal to 4.0 meq/L.
19. Concomitant medications that are potent inducers (rifampicin, rifabutin, phenytoin, carbamazepine, phenobarbital and St. John's Wort) of CYP3A4 function.
20. Hypertension not controlled by medical therapy (systolic blood pressure greater than 160 mm Hg or diastolic blood pressure greater than 100 mm Hg)
21. Presence of left bundle branch block (LBBB.)
22. Any unresolved toxicity greater than common terminology criteria (CTC) grade 1 from previous anti-cancer therapy.
23. Currently active diarrhea that may affect the ability of the patient to absorb the ZD6474 or tolerate diarrhea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne S. Tsao, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Tam AL, Kim ES, Lee JJ, Ensor JE, Hicks ME, Tang X, Blumenschein GR, Alden CM, Erasmus JJ, Tsao A, Lippman SM, Hong WK, Wistuba II, Gupta S. Feasibility of image-guided transthoracic core-needle biopsy in the BATTLE lung trial. J Thorac Oncol. 2013 Apr;8(4):436-42. doi: 10.1097/JTO.0b013e318287c91e. PMID 23442309
- [Derived] Kim ES, Herbst RS, Wistuba II, Lee JJ, Blumenschein GR Jr, Tsao A, Stewart DJ, Hicks ME, Erasmus J Jr, Gupta S, Alden CM, Liu S, Tang X, Khuri FR, Tran HT, Johnson BE, Heymach JV, Mao L, Fossella F, Kies MS, Papadimitrakopoulou V, Davis SE, Lippman SM, Hong WK. The BATTLE trial: personalizing therapy for lung cancer. Cancer Discov. 2011 Jun;1(1):44-53. doi: 10.1158/2159-8274.CD-10-0010. Epub 2011 Jun 1. PMID 22586319
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: November 2006 to February 2010. All participants recruited at The University of Texas MD Anderson Cancer Center.
Groups:
- ZD6474: ZD6474 300 mg by mouth daily.
Period: Overall Study
Arm/Group | ZD6474
Started | 54
Completed | 54
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ZD6474
Number analyzed (Participants) | 54
Age, Continuous [Mean (Full Range); unit: years] | 61 [34 to 80]
Age, Customized [Number; unit: participants]
  <=50 years | 11
  Between 51 and 60 years | 15
  Between 61 and 70 years | 19
  >70 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 54

OUTCOME MEASURES:

1. Secondary Outcome: 8 Week Progression-Free Survival
Description: Progression-free survival (PFS) was estimated using Kaplan-Meier method. PFS was defined as time from start of treatment to disease progression.
Time Frame: Every 8 weeks till disease progression.
Measure: Median (Full Range); unit: months
Arm/Group | ZD6474
Number analyzed (Participants) | 54
months | 1.81 [0.16 to 23.46]

2. Primary Outcome: 8-Week Disease Control Rate (Complete Response, Partial Response and Stable Disease)
Description: The disease control rate (DCR) is the percentage of patients without progression at 8 weeks. Disease control rate defined as: Complete Response (CR): Disappearance of all non-target/target lesions and normalization of tumor marker level. Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum LD since the treatment started.
Time Frame: Baseline to 8 Weeks
Measure: Number; unit: percentage of participants
Arm/Group | ZD6474
Number analyzed (Participants) | 54
percentage of participants | 33

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were assessed from the time of consent until 30 days following the last dose of study treatment.
Description: Collection period: January 16, 2007 to April 02, 2010.
Arm/Group | ZD6474
Serious Adverse Events (participants affected / at risk) | 54/54
Other Adverse Events (participants affected / at risk) | 54/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZD6474 (N=54)
Febrile Neutropenia (Infections and infestations) | 6 (6)
Respiratory Infection (Infections and infestations) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Lipase Abnormal (Metabolism and nutrition disorders) | 2 (2)
Multifold Ischemic Disease of CNS (Vascular disorders) | 1 (1) — CNS - Central Nervous System
Skin Hemorrhage (Skin and subcutaneous tissue disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Large Intestine Perforation (Gastrointestinal disorders) | 2 (2)
Blood Creatinine Increased (Blood and lymphatic system disorders) | 5 (5)
Acute Renal Failure (Renal and urinary disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiorespiratory Arrest (Cardiac disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 4 (4)
Hypoalbuminemia (Hepatobiliary disorders) | 1 (1)
Neutropenia (Infections and infestations) | 8 (8)
Dysgeusia (Gastrointestinal disorders) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Oesophageal Varices Hemorrhage (Gastrointestinal disorders) | 1 (1)
Bronchitis Bacterial (Infections and infestations) | 1 (1)
Perforated Right Cornea (Eye disorders) | 1 (1)
Intestinal Perforation (Gastrointestinal disorders) | 5 (5)
Depressed Level of Consciousness (Nervous system disorders) | 4 (4)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 5 (5)
Cardiac Failure (Cardiac disorders) | 1 (1)
Gastric Ulcer (Gastrointestinal disorders) | 2 (2)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Hypertension (Cardiac disorders) | 2 (2)
Cerebral Hemorrhage (Cardiac disorders) | 4 (4)
Hematocrit Decreased (Blood and lymphatic system disorders) | 1 (1)
Gait Distrubance (Musculoskeletal and connective tissue disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Opportunistic Infection (Infections and infestations) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (General disorders) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 4 (4)
Rectal Hemorrhage (Gastrointestinal disorders) | 1 (1)
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemorrhage (Blood and lymphatic system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Pyramidal Tract Syndrome (Nervous system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 4 (4)
Septic Shock (Infections and infestations) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Death (General disorders) | 10 (10)
Papilloedema (Vascular disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Peripheral Sensorimotor Neuropathy (Nervous system disorders) | 2 (2)
Retinal Artery Occlusion (Vascular disorders) | 1 (1)
Appendicitis (Gastrointestinal disorders) | 2 (2)
Convulsion (Musculoskeletal and connective tissue disorders) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Pancreatitis (Hepatobiliary disorders) | 1 (1)
Purulent Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Peripheral Motor Neuropathy (Nervous system disorders) | 1 (1)
Thromboplastin (Blood and lymphatic system disorders) | 1 (1)
Infection (Infections and infestations) | 4 (4)
Post Operative Wound Infection (Infections and infestations) | 1 (1)
Intestinal Infection (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cognitive Disorder (Psychiatric disorders) | 1 (1)
Cardiac Troponin (Cardiac disorders) | 1 (1)
Bartholin Abscess (Infections and infestations) | 1 (1)
Perforated Diverticulum (Gastrointestinal disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Hemoptysis (Blood and lymphatic system disorders) | 1 (1)
Chest Pain (General disorders) | 3 (3)
Acute Respiratory Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 2 (2)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 1 (1)
Tumor Hemorrhage (Blood and lymphatic system disorders) | 2 (2)
Enterovesical Fistula (Gastrointestinal disorders) | 2 (2)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Thrombolysis (Blood and lymphatic system disorders) | 1 (1)
Pulmonary Edema (Cardiac disorders) | 1 (1)
Sepsis (Immune system disorders) | 1 (1)
Edema Peripheral (General disorders) | 1 (1)
Enterocutaneous Fistula (Gastrointestinal disorders) | 1 (1)
Proctorrhagia (Gastrointestinal disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Gallbladder Perforation (Hepatobiliary disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
General Physical Health Deterioration (General disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Gamma-glutamyl transferase (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 5 (5)
Pleuropericarditis (Cardiac disorders) | 1 (1)
Anal Fissure (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 2 (2)
Colovesical Fistula (Gastrointestinal disorders) | 1 (1)
Drug Interaction (Investigations) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Diabetic Hyperglycemic Coma (Metabolism and nutrition disorders) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (2)
Vasculitis Cerebral (Vascular disorders) | 1 (1)
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Wound Complication (General disorders) | 1 (1)
Abdominal Perforation (Gastrointestinal disorders) | 1 (1)
PAS Chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Facial Swelling (General disorders) | 1 (1)
Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lymphocyte Count Decreased (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZD6474 (N=54)
Abnormal Electrolytes (Renal and urinary disorders) | 25 (25)
Constitutional Symptoms (General disorders) | 24 (24)
Diarrhea (Gastrointestinal disorders) | 24 (24)
Elevated Alkaline Phosphatase (Metabolism and nutrition disorders) | 22 (22)
Abnormal Liver Enzymes (Hepatobiliary disorders) | 19 (19)
Hypertension (Cardiac disorders) | 18 (18)
Rash (Skin and subcutaneous tissue disorders) | 11 (11)
Anorexia (Gastrointestinal disorders) | 15 (15)
Hyperglycemia (Metabolism and nutrition disorders) | 15 (15)
Pain (General disorders) | 5 (5)
Proteinuria (Metabolism and nutrition disorders) | 14 (14)
Gastrointestinal Complaint (Gastrointestinal disorders) | 13 (13)
Infection (Infections and infestations) | 1 (1)
Renal Insufficiency (Renal and urinary disorders) | 12 (12)
Anemia (Blood and lymphatic system disorders) | 14 (14)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Bleed (Blood and lymphatic system disorders) | 10 (10)
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 (10)
Abdominal Bloating (Gastrointestinal disorders) | 1 (1)
Abdominal Cramps (Gastrointestinal disorders) | 1 (1)
Allergies (General disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Arrythmia, Tachycardia (Cardiac disorders) | 1 (1)
Arrythmia,PAC's (Cardiac disorders) | 1 (1)
Arrythmia,Tachycardia (Cardiac disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Bleeding Gums (Blood and lymphatic system disorders) | 1 (1)
Brusing (Skin and subcutaneous tissue disorders) | 1 (1)
Cardiac Ischemic (Cardiac disorders) | 1 (1)
Central Nervous System Hemorrhage (Nervous system disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Constitutional Cold Sensitive (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Decreased Chloride (Metabolism and nutrition disorders) | 1 (1)
Decreased GFR (Renal and urinary disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 2 (2)
Dehydration (General disorders) | 2 (2)
Depression (Nervous system disorders) | 2 (2)
Diplopia (Eye disorders) | 1 (1)
Dizziness (Nervous system disorders) | 6 (6)
Dry Eye Syndrome (Eye disorders) | 2 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 4 (4)
Dysgeusia (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Dysphasia (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Dysuria (Renal and urinary disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Edema, Bilateral Ankles (Blood and lymphatic system disorders) | 1 (1)
Edema, Left Neck (Blood and lymphatic system disorders) | 1 (1)
Elevated Troponin (Cardiac disorders) | 1 (1)
Elevated ALT (Metabolism and nutrition disorders) | 16 (16)
Elevated Amylase (Metabolism and nutrition disorders) | 1 (1)
Elevated AST (Metabolism and nutrition disorders) | 17 (17)
Elevated Creatine (Metabolism and nutrition disorders) | 1 (1)
Elevated Creatinine (Metabolism and nutrition disorders) | 11 (11)
Elevated Glucose (Metabolism and nutrition disorders) | 3 (3)
Elevated INR (Blood and lymphatic system disorders) | 1 (1)
Elevated Lipase (Metabolism and nutrition disorders) | 1 (1)
Elevated Prothrombin Time (Blood and lymphatic system disorders) | 4 (4)
Elevated Partial Thromboplastin Time (Blood and lymphatic system disorders) | 4 (4)
Elevated WBC (Blood and lymphatic system disorders) | 6 (6)
Epistaxis (General disorders) | 2 (2)
Fatigue (General disorders) | 20 (20)
Fever (General disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hemoglobinuria (Metabolism and nutrition disorders) | 3 (3)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hot Flashes (Endocrine disorders) | 1 (1)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 4 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 7 (7)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 6 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (7)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 5 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 9 (9)
Hyponatremia (Metabolism and nutrition disorders) | 12 (12)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3)
Hypotension (Cardiac disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection, Ear (Infections and infestations) | 1 (1)
Infection, Eyes (Infections and infestations) | 1 (1)
Infection, Respiratory (Infections and infestations) | 1 (1)
Infection, Toenail (Infections and infestations) | 2 (2)
Insomnia (General disorders) | 1 (1)
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 3 (3)
Lymphopenia (Infections and infestations) | 2 (2)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (8)
Neuropathy (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain, Abdominal (Gastrointestinal disorders) | 3 (3)
Pain, Back (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain, Chest (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain, Heel (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, Left Knee and Shin (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, Left Scapula (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, Lumbar (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, Right Ear (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, Right Foot (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, Right Side (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, Waist to Shoulder (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, Right Arm (Musculoskeletal and connective tissue disorders) | 1 (1)
Pelvic Ascites (Gastrointestinal disorders) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Progression of Disease NOS (General disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
QTC Prolongation (Cardiac disorders) | 5 (5)
Rash, Acneiform (Skin and subcutaneous tissue disorders) | 5 (5)
Rash, Chest (Skin and subcutaneous tissue disorders) | 1 (1)
Rash, Pubic Area (Skin and subcutaneous tissue disorders) | 1 (1)
Rash, Hands (Skin and subcutaneous tissue disorders) | 3 (3)
Seizures (Nervous system disorders) | 3 (3)
Sepsis (Immune system disorders) | 1 (1)
Severe Aortic Insufficiency (Cardiac disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Stomatitis (Infections and infestations) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Tooth Abscess (Infections and infestations) | 1 (1)
Tremors (Nervous system disorders) | 2 (2)
Unsteady Gait (Musculoskeletal and connective tissue disorders) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 6 (6)
Vision Floaters (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5)
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Weight Loss (General disorders) | 5 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Xerostomia (Gastrointestinal disorders) | 1 (1)
Rash, Face (Skin and subcutaneous tissue disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No